CLINICAL TRIAL: NCT00394043
Title: Treatment Efficacy of OMT for Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: Osteopathic Research Center (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R21AT002303-01A2 (NIH)
Record Dates: First submitted 2006-10-27; First posted 2006-10-31 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Sydrome; Osteopathic Manipulative Treatment; Osteopathic Manipulative Medicine; Physical Medicine
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Osteopathic Manipulative Treatment (Experimental): A protocol of specific osteopathic manipulative techniques was applied.
  Interventions: Procedure: Osteopathic Manipulative Treatment
- Placebo ultrasound (Placebo Comparator): Sub-therapeutic ultrasound was applied.
  Interventions: Procedure: Placebo Sub-Therapeutic Ultrasound
- Standard Medical care (No Intervention): Subjects did not receive either study treatment, but continued to receive standard medical care.

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — A protocol of specific Osteopathic manipulative techniques was used.
  Arms: Osteopathic Manipulative Treatment
Procedure: Placebo Sub-Therapeutic Ultrasound — Sub-therapeutic ultrasound was applied in a standardized method.
  Arms: Placebo ultrasound

SUMMARY:
This study investigated whether an eight-week regimen of osteopathic manipulative treatment would have immediate and lasting positive effects on the symptoms, functional limitation and physiologic impairment associated with Carpal Tunnel Syndrome.

DETAILED DESCRIPTION:
The incidence of Carpal Tunnel Syndrome (CTS) in adults in the U.S. ranges from 15-20% depending on the study, and costs over one billion dollars annually in medical care. Surgery for CTS accounts for much of these costs with up to one third of these patients experiencing re-occurrence of symptoms post-operatively.

The overall goal for this proposed exploratory clinical trial was to evaluate the efficacy of a conservative, manual medicine treatment as an adjunctive therapy to standard care for CTS. This pilot study utilized a prospective, randomized, placebo-controlled clinical trial methodology to examine whether an eight week treatment regimen of osteopathic manipulative treatment (OMT) when used adjunctively to standard therapy would have immediate and lasting positive effects on the symptoms, functional limitations, and physiologic impairment associated with CTS.

Male and female subjects between the ages of 20 and 65 who meet electro-physiologic and symptom/functional inclusion criteria were randomly assigned to one of three study groups, all of which will continue standard medical care with their treating physician/provider; (i) OMT plus standard medical care; (ii) placebo (sub-therapeutic ultrasound) plus standard medical care; and (iii) standard medical care only (no-treat).

Outcome measures were: 1. Median and Ulnar motor and sensory nerve conduction amplitudes and distal latencies, 2. Symptoms and Functional status, 3. Strength, 4. Sensation, 5. Interior dimensions of the carpal tunnel, and 6. Quantification (signal intensity by MRI) of water (edema) in the Median nerve and carpal tunnel. Placebo potency and blinding success will be evaluated. A preliminary investigation demonstrated our ability to recruit subjects and measure these outcomes. Power analysis based upon a decrease in the mean median motor nerve distal latency of 30% identified a minimum number of 42 subjects per treatment group.

It was expected that a significantly greater number of subjects in the OMT adjunctive treatment group would achieve the effective change in nerve latency compared to the other two treatment groups. It was also expected that the OMT adjunctive treatment group would have greater improvement of all physiological and clinical outcome measures than the other two groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with a self-reported medical diagnosis of unilateral or bilateral CTS, between the ages of 21 and 65 and all races and ethnic groups.
* Median motor nerve distal latency greater than 4.2 ms
* A difference between ipsilateral Median and Ulnar motor nerve distal latency greater than 1.5 ms.
* Median nerve sensory nerve distal latency greater than 2.2 ms
* A difference between Median and Ulnar sensory nerve peak distal latency greater than 0.2 ms

Exclusion Criteria:

* severe CTS that has progressed to muscle atrophy
* pregnancy
* previous wrist surgery on the wrist to be studied
* systemic disease or condition including but not limited to diabetes mellitus, thyroid disorders, rheumatoid disorders, Paget's bone disease, gout, myxedema, multiple myeloma, acromegaly, hepatic disease, dialysis patients, or other diseases or conditions in which peripheral neuropathies are common.
* secondary cause of CTS such as a ganglion cyst, mass, or an accessory muscle shown by an MRI exam of the wrist.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Changes in the Median motor and sensory distal latencies.
Improvement in the patients'self-reported symptoms and functionality scores.

SECONDARY OUTCOMES:
Strength measured with one grip and three pinch strength tests.
Changes in sensation as measured by Current Perceptual Threshold.
Changes in the transverse and anterior/posterior interior diameters and cross-sectional areas of the carpal tunnel.
Carpal tunnel edema.

CONTACTS AND LOCATIONS:
Overall Officials: Scott T Stoll, D.O., Ph.D., Principal Investigator — Osteopathic Research Center University of North Texas Health Science Center